CLINICAL TRIAL: NCT05166473
Title: Are Telerehabilitation Exercise Practices Effective In Patients Diagnosed With Beign Paroxysmal Positional Vertigo?
Brief Title: Effectiveness of Telerehabilitation Exercise for Bening Paroxysmal Positional Vertigo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alanya Alaaddin Keykubat University (Other)
Responsible Party: Principal Investigator, Ayça Araci, Physical Therapist,principal investigator, pHd, Alanya Alaaddin Keykubat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10354421-2021/07-09
Record Dates: First submitted 2021-09-07; First posted 2021-12-22 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Benign Paroxysmal Vertigo
Keywords: Bening paroxysmal vertigo; telerehabilitation; physiotherapy; halpike maneuver; exercise
MeSH Terms: conditions — Motor Activity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant
Masking Description: it was calculated that 80% power could be achieved in the 95% confidence December when at least 42 people (at least 21 people for each group) were taken into the study. In all tests, the statistical significance level was taken as p<0.05.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (n=21) (Experimental): This group was conducted with a physiotherapist for video conference-based vestibular rehabilitation exercises, was called the "telerehabilitation group (TR)". In terms of ease of Use and applicability, the WhatsApp app was preferred. Patients were individually searched for two days a week, 25-30 minutes. The exercises were performed gradually from easy to difficult, initially in a sitting position in accordance with the levels of the patients.
  Interventions: Other: Telerehabilitation group (n=21)
- Control Group (n=21) (Active Comparator): After the home exercise program, which should be applied twice a day for six weeks, was shown in practice, the home exercise program was given, in which the exercises were visual and written, this group was called the "control group". All participants were given a phone number to consult when there were any problems, and were phoned to decry whether they were continuing the exercises.
  Interventions: Other: Control Group (n=21)

INTERVENTIONS:
Other: Telerehabilitation group (n=21) — This group was conducted with a physiotherapist for video conference-based vestibular rehabilitation exercises, was called the "telerehabilitation group (TR)". In terms of ease of Use and applicability, the WhatsApp app was preferred. Patients were individually searched for two days a week, 25-30 minutes. The exercises were performed gradually from easy to difficult, initially in a sitting position in accordance with the levels of the patients.
  Arms: Telerehabilitation group (n=21)
Other: Control Group (n=21) — After the home exercise program, which should be applied twice a day for six weeks, was shown in practice, the home exercise program was given, in which the exercises were visual and written, this group was called the "control group". All participants were given a phone number to consult when there were any problems, and were phoned to decry whether they were continuing the exercises.
  Arms: Control Group (n=21)

SUMMARY:
In addition to the channelize reposition maneuvers (KRM) that will be applied by the physician in patients diagnosed with Benign paroxysmal positional Vertigo (BPPV), the aim of the study is to investigate the effect of vestibular rehabilitation exercises that will be October based on telerehabilitation by the physiotherapist.

DETAILED DESCRIPTION:
Benign paroxysmal positional vertigo (BPPV), the most common form of recurrent vertigo the common cause. Short-term, occurring with specific head movements, it is described as episodic, transient vertigo attacks.Calcium in the movement of the head autocoids formed from carbonate crystals emerge from the places and one or more crystals enter the semicircular channel, which affects the endolymphatic flow of the Vertigo leads to the formation. BPPV is also characterized by positional nystagmus along side positional vertigo. BPPV often causes a person to restrict person's life and weeks or it recovers spontaneously within months. Autolytic debrides in the cupula aimed at separating the cupula or removing the clutches from the canal vestibular exercises or maneuvers significantly accelerate healing. In the treatment of BPPV, vestibular rehabilitation applications are used primarily.As a vestibular rehabilitation, the canalith reposition maneuver, developed by Epley and effective, is often preferred. Telerehabilitation, rehabilitation by the use of electronic communication systems describes the provision of services to patients remotely. Transport to health services to provide an effective rehabilitation service to patients when limited it takes advantage of telerehabilitation. Some studies show that telerehabilitation can reduce health care costs, improve physical and mental function and quality of life, and be presented in a way that satisfies patients.The Covid-19 epidemic outbreak has affected health care. To protect healthcare workers and patients from the risk of infection, to ensure widespread use of telecommunications technology instead of face-to-face clinical visits, rules, regulations.With these arrangements, telerehabilitation became of great importance for physiotherapists.High levels of evidence on image-based telerehabilitation technologies suggest that they can be used for remote diagnosis and patient follow-up and are the most effective method for physiotherapists. Pain of exercise through telerehabilitation compared to other interventions, it has at least similar effects on physical function and quality of life references. As a method of vestibular rehabilitation, mostly when examined in the literature it has been observed that manoeuvring has been applied and these practices have been compared with drugs. In this study, aim is to support the literature by adding exercise practices given according to the levels of telerehabilitation-based patients along with maneuver practices.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with positional vertigo,
* Be in the December 18-65 age range
* Dix Hallpike maneuver test ( + ),
* Who volunteers to participate in the study
* Sufficient to use technology,
* Can understand the instructions given in Turkish
* Having smart phone and active internet connection

Exclusion Criteria:

* At the end of the examination, there are signs of acute or chronic infection
* Thought to have neurological pathology that causes dizziness
* Head trauma, with a history of surgical operation
* Lower extremity pain that prevents you from standing and giving a load
* A history or symptom of diseases of the vestibular system other than BPPV
* Lower limb surgery
* Sudden sensorial hearing loss and the presence of chronic otitis media

  • Pregnancy
* Presence of a serious cognitive disorder detected by a doctor at a level that will prevent testing
* Not being at a mental level to understand and answer survey questions
* Cervical pathologies that can lead to dizziness

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Tandem test | "baseline" and "immediately after the intervention"
  The patient positioned the heel of one foot so that it came to the tip of the finger of the other foot. He tried to maintain his position for 30 seconds with his hands outstretched and eyes open and closed in parallel. Duration recorded in sec.
Change in Semitandem test | "baseline,preintervention " and "immediately after the intervention"
  The patient positioned his feet so that one foot was slightly in front of and adjacent to the other. He tried to maintain his position for 30 seconds with his hands outstretched and eyes open and closed in parallel. The length of time it could stop was recorded in second.
Change in Dizziness disability inventory (BEE) score: | "baseline" and "immediately after the intervention"
  It provides the determination of the factors that cause dizziness and balance disorder of patients experiencing dizziness and their physical, functional and sensory status in diseases of the vestibular system.The inventory consists of 25 questions. It contains 7 questions that study physical effects, 9 questions that study functional effect, and 9 questions that include emotional factors. The answers to the questions are given yes (4 points) , sometimes (2 points), no (0 points). The maximum score of the factors studying physical effects is 28, the maximum score of the factors studying sensory and functional effects is 36 points. A high score indicates that a person has high symptoms of dizziness, and dizziness is considered to cause restriction in their daily life activities.
Change in Vertigo symptom scale | "baseline" and "immediately after the intervention"
  Vertigo symptom scale is a scale designed to determine somatic anxiety and autonomic complaint in patients with dizziness complaints.It contains 8 articles related to vertigo (0-32 points), 7 articles containing autonomic complaints (0-28 points).
Change in Beck anxiety scale | "baseline" and "immediately after the intervention"
  The Beck Anxiety Scale was used to determine patients ' anxiety levels and frequency of symptoms.0 points: none, 1 point: light , 2 points: medium , 3 points: seriously determined. (8-15 points ) mild anxiety symptoms are defined as moderate (16-25 points), moderate (26-63 points), severe anxiety level.
Change in Vertigo Dizziness Imbalance Questionnaire | "baseline" and "immediately after the intervention"
  It is used to measure the frequency of vertigo and dizziness complaints in patients and to determine how much their quality of life is affected.It consists of 14 questions for symptoms and 22 questions for measuring the quality of life. In the survey, which contains a total of 36 questions, the questions are scored as 0: all the time, 1: most of the time, 2: often, 3: sometimes, 4: very infrequently and 5: never. The total score on the symptom scale is 70, and the quality of life is 100. The high score obtained indicates that the person has few symptoms and has a high quality of life.
Chang in Visual Analog Scale | "baseline" and "immediately after the intervention"
  The Visual Analog scale (VAS) has been used to determine the severity of dizziness. The patient is asked to score between 0 and 10.0: I don't have dizziness, 1-4: Mild severity, 4-8: Moderate severity, 10: I have unbearable dizziness.
Change in Romberg test | "baseline" and "immediately after the intervention"
  When the patients stand in a correct posture, postural control is provided by visual, somatosensory, vestibular system stimuli. In the Romberg test, the patient stood with the feet united. He joined his hands diagonally in front of the trunk. He tried to maintain his position for 30 seconds with his eyes closed. If there is a disorder of the vestibular system, the patient has a tendency to fall towards the side where the lesion is located.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Alanya Alaaddin Keykubat Üniversity, Antalya, Alanya
  - Alanyaaku, Antalya, Alanya

IPD SHARING:
Plan to Share IPD: No